CLINICAL TRIAL: NCT01907776
Title: A Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of ME1100 Inhalation Solution (Arbekacin Inhalation Solution) Administered to Healthy Volunteers
Brief Title: Pharmacokinetics and Safety Study of ME1100 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Meiji Seika Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ME1100-CL-101
Record Dates: First submitted 2013-07-22; First posted 2013-07-25 (Estimated); Last update posted 2014-06-12 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
MeSH Terms: interventions — arbekacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ME1100 (Experimental): ME1100 inhalation solution (arbekacin for oral inhalation at 150 mg/mL), 0.6, 2.0, 3.0, 4.0, 6.0, or 9.0mL, Single Dose
  Interventions: Drug: ME1100 inhalation solution
- Placebo (Placebo Comparator): ME1100 placebo inhalation solution
  Interventions: Drug: ME1100 placebo inhalation solution

INTERVENTIONS:
Drug: ME1100 inhalation solution — ME1100 inhalation solution (arbekacin for oral inhalation at 150mg/mL), 0.6, 2.0, 3.0, 4.0, 6.0, or 9.0mL, Single Dose
  Other Names: arbekacin; ME1100
  Arms: ME1100
Drug: ME1100 placebo inhalation solution — Vehicle placebo
  Arms: Placebo

SUMMARY:
This is a single-center, randomized, double-blind, placebo-controlled, sequential group study. The primary objective of this study is to assess the tolerability and safety of single doses of ME1100 inhalation solution (orally inhaled arbekacin). The secondary objective is to determine the systemic exposure to, and urinary elimination of, ME1100.

ELIGIBILITY:
Inclusion Criteria:

* Male (who are surgically sterile or agree to practice barrier contraception throughout their participation in the study) or Female (using oral or double barrier contraceptive if sexually active, surgically sterile or post-menopausal confirmed by follicle stimulation hormone test);
* Willing to give written informed consent
* 18 to 55 years of age at time of consent
* Body Mass Index of 18-30 kg/m2
* Non-smoker (for at least 6 months prior to screening) and willing to abstain from smoking during the course of the study
* Good general health as determined by medical history, physical examination, 12-lead electrocardiograms and clinical laboratory tests (including normal renal function and high frequency audiometry)
* Willing to abstain from alcohol, caffeine, and xanthine-containing beverages for 24 hours prior to and 72 hours after dosing.
* Japanese subjects must be first generation Japanese (4 grandparents, biologic parents and subject born in Japan)

Exclusion Criteria:

* Uncontrolled, clinically significant disease which in the opinion of the Principal Investigator or Medical Monitor would place the subject at risk through study participation or would confound the assessment of the safety of ME1100 inhalation solution
* Evidence of current or history of respiratory disease, including asthma, emphysema, chronic bronchitis, or cystic fibrosis
* History or current symptom(s) of respiratory tract inflammation within 30 days of Visit 2
* History of hearing, balance or ear disorder or surgery or injury to the ears, or with genetic mutation (>5.0% heteroplasmy) suggestive of increased risk of hearing loss (MT-RNR1 [A1555G] for mitochondrial 12S ribosomal RNA gene or MT-TS1 [A3243G] for mitochondrial transfer RNA serine 1)
* History of parent, sibling or parental sibling reporting hearing loss before age 65 years
* History of malignancy
* History of clinically significant alcohol or drug abuse
* History within last 6 months or current use of any tobacco product including e-cigarettes
* Positive drug screen for drugs of abuse
* Positive test for HIV, Hepatitis B or Hepatitis C
* Use of any prescription or over-the-counter medications (except oral or hormonal contraceptives), herbal supplements, or vitamins within 14 days of Visit 2
* Known hypersensitivity to any aminoglycoside or bacitracin antibiotic
* Female of childbearing potential with a positive urine pregnancy test, or currently breast feeding.
* Inability to perform reproducible spirometry in accordance with American Thoracic Society (ATS) guidelines
* Abnormal Forced Expiratory Volume in the First Second (FEV1), Forced Vital Capacity (FVC), or FEV1/FVC (FEV1 or FVC < 80% of predicted or FEV1/FVC ratio < 0.7)
* FEV1 variability > 10% between Visit 1 and Visit 2 (prior to dosing)
* Significant blood donation (or testing) in previous 8 weeks before screening.
* Use of any Investigational Product in previous 30 days or 5 half-lives, whichever is longer, preceding start of screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2013-07; Primary Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | from Baseline to Day 8-10
Number of participants with abnormal physical examinations | from Baseline to Day 8-10
Number of participants with abnormal 12-lead electrocardiograms | from Baseline to Day 8-10
Number of participants with abnormal vital signs | from Baseline to Day 8-10
Number of participants with abnormal safety laboratory measurements | from Baseline to Day 8-10

SECONDARY OUTCOMES:
Serum Concentration of ME1100 | 5, 15, 30 minutes and 1, 2, 3, 4, 6, 8, 12, 18 and 24 hours post START of dosing
Urinary elimination of ME1100 | 0-6, 6-12, 12-24, 24-48 and 48-72 hours after single dosing

CONTACTS AND LOCATIONS:
Overall Officials: Mitsuharu Egawa, Study Chair — Meiji Seika Pharma Co., Ltd.
Locations (1):
- WCCT Global, LLC, Cypress, California, United States